CLINICAL TRIAL: NCT07240792
Title: Expanding Mental Health Access in Rural High Schools: Development and Testing of a College Student-Delivered Cognitive-Behavioral Therapy (CBT) Intervention
Brief Title: Development of a College Student-Delivered Cognitive-Behavioral Therapy (CBT) Intervention for Rural High School Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jamal Essayli, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27316
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Depression; Anxiety; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Student Delivered Cognitive Behavioral Therapy (CBT) Intervention (Experimental): The investigators will develop an intervention protocol drawing from evidence-based cognitive-behavioral therapy (CBT) components, including psychoeducation, behavioral activation, exposure therapy, cognitive restructuring, and problem solving, tailored to address the mental health needs in rural high school students and implemented by undergraduate college students.
  Interventions: Behavioral: Student Delivered Cognitive Behavioral Therapy Intervention

INTERVENTIONS:
Behavioral: Student Delivered Cognitive Behavioral Therapy Intervention — Our study aims to evaluate whether a 12-week cognitive-behavioral therapy (CBT) program delivered in both group and individual formats by trained college students can effectively help adolescents with symptoms of depression, anxiety, and stress. We will assess the program's feasibility, acceptability, and effectiveness in a high school setting. Sessions will cover topics such as: understanding connections between thoughts, feelings, and behaviors, identifying and challenging unhelpful thought patterns, using exposure principles to face feared situations, building problem-solving skills, and engaging in positive activities.

SUMMARY:
This research is being done to find out the effectiveness, feasibility, and acceptability of a college student-delivered cognitive-behavioral therapy (CBT) intervention in high schools in rural Schuylkill County, Pennsylvania to treat mental health problems (i.e. depression and anxiety) in adolescents. This project will respond to the need for evidence-based, acceptable, accessible, and low-cost adolescent cognitive-behavioral interventions that lead to long-term improvements in adolescents' mental health outcomes.

DETAILED DESCRIPTION:
The overarching goal of this study is to iteratively adapt and test an innovative mental health delivery model that leverages college students to provide cognitive-behavioral therapy (CBT) to high school students in rural Schuylkill County, Pennsylvania. The investigators' preliminary data and established Community Advisory Board (CAB) support three key premises that drive this project. First, depression, anxiety, and stress are the most prevalent mental health challenges facing rural adolescents. Second, multiple barriers impede access to mental health care in rural communities, including provider shortages, mental health stigma, cost, insurance constraints, and limited parental knowledge or support. Third, these barriers can be addressed by enhancing school-based mental health services through a novel delivery model: licensed psychologists training undergraduate students to provide CBT interventions directly in high school settings.

Aim 1: Iteratively adapt and pilot CBT for high school students in rural Pennsylvania. The investigators will employ a systematic adaptation process guided by their preliminary data and the Framework for Reporting Adaptations and Modifications-Enhanced (FRAME) to develop a culturally responsive and contextually appropriate CBT intervention for rural high school settings. This iterative refinement process will integrate feedback from two complementary sources: (1) semi-structured interviews with high school student participants and college student interventionists; and (2) a CAB comprising high school students, parents/caregivers, school mental health providers, school administrators, and college student interventionists. By the end of the two-year project period, the investigators will have developed a CBT intervention specifically tailored for high school students in rural Pennsylvania, with clear documentation of adaptation decisions and their empirical basis.

Aim 2: Examine the effects of the adapted CBT intervention on mental health outcomes among rural high school students. The investigators will evaluate preliminary effectiveness using self-report measures of depression, anxiety, and stress in 24-40 high school students (6-10 students/CBT group) across four implementation periods. Outcomes will be measured at pre-treatment, mid-treatment, and post-treatment. The investigators hypothesize that the adapted CBT intervention will result in at least a 50% decrease in mental health symptoms.

Aim 3: Evaluate the feasibility, acceptability, engagement, and fidelity of the adapted CBT intervention. The investigators will employ a mixed-methods approach to comprehensively evaluate four key implementation outcomes. Feasibility will be assessed through recruitment and retention metrics, while acceptability will be measured via standardized instruments and stakeholder feedback. Engagement will be tracked through session attendance and participation rates, and fidelity will be monitored through systematic assessment of intervention delivery. The investigators hypothesize that the adapted CBT intervention will meet or exceed pre-determined benchmarks across all implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* High school students ages 13-18 years.
* Attending a participating rural high school in Schuylkill County, Pennsylvania.
* Presenting with self-reported symptoms of depression, anxiety, or stress. Must have a t-score ≥ 55 on one or more of the following three measures:

  i. PROMIS Emotional Distress Depression short-form questionnaire ii. PROMIS Emotional Distress Anxiety short-form questionnaire iii. PROMIS Psychological Stress Experiences short-form questionnaire
* English-speaking (to ensure comprehension of CBT materials and assessments).

Exclusion Criteria:

* Diagnosis of a psychotic disorder, bipolar disorder, intellectual disability, or seizure disorder.
* Assessed to be at high risk for suicide or requiring immediate crisis intervention.
* Inability to participate in school-based sessions due to scheduling conflicts or behavioral concerns.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) 8-item Emotional Distress-Depression | Baseline, Week 6, Week 12
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression measure is an 8-item self-report questionnaire that examines depressive symptoms. Scores range from 8-40, with higher scores indicating higher levels of depression.
PROMIS 8-item Emotional Distress-Anxiety | Baseline, Week 6, Week 12
  The PROMIS Emotional Distress-Anxiety measure is an 8-item self-report questionnaire that examines anxiety symptoms. Scores range from 8-40, with higher scores indicating higher levels of anxiety.
PROMIS 8-item Psychological Stress Experiences | Baseline, Week 6, Week 12
  The PROMIS Psychological Stress Experiences measure is an 8-item self-report questionnaire that examines stress symptoms. Scores range from 8-40, with higher scores indicating higher levels of stress.
Recruitment Rate | Through study completion, an average of 2 years
  The investigators will determine the percent of participants recruited who consented to the study and attended the initial session.
Retention Rate | Through study completion, an average of 2 years
  The investigators will determine the percent of participants consented who completed all study measures.

SECONDARY OUTCOMES:
Participant Engagement | Through study completion, an average of 2 years
  The investigators will measure engagement through session attendance rates and session participation tracking.
Credibility/Expectancy Questionnaire (CEQ) | Week 6, Week 12
  The Credibility/Expectancy Questionnaire (CEQ) is a 6-item questionnaire that examines the participants' perceptions of treatment credibility and their expectations for improvement. Scores range from 4-36 for questions 1, 2, 3, and 5. Questions 4 and 6 use a 0-100% scale. Higher scores indicate a more positive perception of the treatment and lower scores indicate a more negative perception of the treatment.
Intervention Fidelity | Through study completion, an average of 2 years
  The investigators will measure intervention fidelity via systematic fidelity monitoring through an adapted CBT checklist completed by interventionists after each session. A random sample of sessions (20%) will be audio-recorded and rated by independent evaluators to verify self-reported fidelity.